CLINICAL TRIAL: NCT06786663
Title: Feasibility Study for the Generation of Organoids From Male Breast Tumors
Brief Title: MALE Mamm Organoids
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: San Giovanni Addolorata Hospital (Other); Weizmann Institute of Science, Israel (Unknown); S. Andrea Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RS83/IRE/23
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Breast Neoplasms, Male
Keywords: Organoids
MeSH Terms: conditions — Breast Neoplasms, Male

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Organoids from male breast tumor tissue collected during surgery (according to standard clinical practice)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is believed that the use of organoids derived from male breast tumors can be of fundamental support for the definition of the molecular mechanisms underlying the onset of the tumor. Furthermore, the development of such preclinical models could be of significant support for the identification of specific personalized and ad hoc therapeutic treatments for male pathology.

DETAILED DESCRIPTION:
The main objective of the project is to set up at least 5 organoid cultures of male breast cancer derived from patients who have undergone surgery. This study will allow to define the success rate in the generation of organoids.

A secondary objective is to verify the correspondence between the organoids generated and the tumor tissue of origin.

In this regard, broad-spectrum molecular investigations will be carried out, such as mutational analysis of DNA through Whole Exome Sequencing (WES), gene expression profiles through RNA sequencing (RNAseq) and small RNA sequencing, proteomic and metabolomic analysis of both the tumors of origin and the cultures of derived organoids (PDO).

Furthermore, to verify the functional correspondence of the organoids with the tumor of origin, in vitro viability tests will be carried out by treating the PDOs with the same drugs administered to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Men aged >18 years
* Patients with histologically confirmed breast cancer with or without synchronous metastases, who will undergo the relevant surgical intervention
* Adequate biological material to be able to carry out the analyses described above
* Signing of the relevant informed consent form

Exclusion Criteria:

not present

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients
Study Population: Male breast cancer (MBC)
Sampling Method: Non-Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2027-04-19 (Estimated); Study Completion 2027-04-19 (Estimated)

PRIMARY OUTCOMES:
Tumor tissue samples collected | 36 months
  Samples of tumor and peri-tumor tissue from the same patient, obtained at the time of surgery for the preparation of organoids to verify the functional correspondence of the organoid cultures obtained from the patients, with the tumors of origin. The organoids will be treated in vitro with doses equivalent to the plasma levels of the drugs administered to the patients, and the viability of the organoids will be assessed through ATPlite assays. Subsequently, the viability data will be compared with the response data of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS National Cancer Institute "Regina Elena", Rome, Italy

IPD SHARING:
Plan to Share IPD: No